CLINICAL TRIAL: NCT06956846
Title: Efficacy of Topical Insuline Drops in Corneal Epithelial Healing Post PRK in Non Diabetic Patients: an Randomized-controlled Trial
Brief Title: Efficacy of Topical Insuline in Corneal Epithelial Healing Post PRK
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hotel Dieu de France Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: CEHDF2402
Record Dates: First submitted 2025-04-25; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Corneal Epithelial Wound Healing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insulin drops (Active Comparator): Eyes receiving eye drops containing human insulin 1U/mL
  Interventions: Drug: insulin eye drops
- Placebo (Placebo Comparator): Eyes only receiving artificial tears
  Interventions: Drug: Artificial tears eye-drops

INTERVENTIONS:
Drug: insulin eye drops — Use of topical insulin eye drops following a standard excimer laser photo-refractive keratecotmy in myopic/astigmatic patients, in order to examine its efficacy in promoting corneal epithelial healing and patient comfort
  Arms: Insulin drops
Drug: Artificial tears eye-drops — The other arm receiving only artificial tears
  Arms: Placebo

SUMMARY:
A prospective randomized double-blind controlled trial will be conducted. The informed consent of each patient will be obtained prior to the procedure.

All patients will undergo a classic PRK procedure

Patients will be instructed to use eye drops blindly in both eyes at a frequency of six times daily:

* In one eye: Insulin drops formulated by combining regular human insulin with artificial tears containing polyethylene glycol (PEG 400) 0,25% at a concentration of 1 unit per milliliter.
* In the other eye: Placebo drops containing only artificial tears. For the double-blind trial, two identical vials will be provided to each patient: one labeled R (for the right eye) and one labeled L (for the left eye). Using the bloc randomization method, the pharmacy will be the only entity aware of the composition of each vial, ensuring that 50% of patients use insulin drops in the right eye and 50% in the left eye.

Every week the drops will be prepared one day prior to the PRK procedure and will be stored in a refrigerator, to be used within one week of their preparation date.

Patients will be examined by two ophthalmology residents on days 2 and 4 post-operatively.

The size of the epithelial defect in both eyes will be measured using the ImageJ software. Thus, the primary outcome of the study is the ulceration closure rate: the smaller the defect, the faster the epithelial healing is.

Additionally, a comparison of subjective symptoms reported by the patient in each eye will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Myopic or astigmatic patient undergoing excimer laser PRK

Exclusion Criteria:

* diabetes mellitus prior ocular surgery ocular surface disease (including dry eye disease, history of herpetic keratitis) previous ocular trauma use of systemic corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-25 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Corneal epithelial healing | From enrollement to day 4 post PRK
  Corneal epithelial defect will be measured ar Day 2 and Day 4 using slit images.

SECONDARY OUTCOMES:
Pain/discomfort | day 4 post PRK
  Subjective patient paint/discomfort scores will be recorded and compared ar day 2 and day 4

CONTACTS AND LOCATIONS:
Locations (1):
- Hotel Dieu de France hospital, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fernandez, MD Alvarado, et al. "3PC-066 Compounding an eye drop formulation of topical insulin for corneal defects refractory to previous treatment: experience in real clinical practice
- [Background] Serrano-Gimenez R, Contreras-Macias E, Garcia-Bernal A, Fobelo-Lozano MJ. Insulin eye drops for treating corneal ulcer in a non-diabetic patient: regarding a case. Farm Hosp. 2020 Oct 6;44(6):297-299. doi: 10.7399/fh.11521. PMID 33156748
- [Background] Diaz-Valle D, Burgos-Blasco B, Gegundez-Fernandez JA, Garcia-Caride S, Puebla-Garcia V, Pena-Urbina P, Benitez-Del-Castillo JM. Topical insulin for refractory persistent corneal epithelial defects. Eur J Ophthalmol. 2021 Sep;31(5):2280-2286. doi: 10.1177/1120672120958307. Epub 2020 Sep 21. PMID 32951459
- [Background] Gómez, M. M., Albaladejo, P. M., Sanz, I. R., Crespo, C. B., Durán, J. P., Alemany, A. L., ... & Martí, M. C. (2022). 3PC-020 Chemical stability and physical compatibility of insulin eye drops used in clinical practice.
- [Background] Castro Mora MP, Palacio Varona J, Perez Riano B, Laverde Cubides C, Rey-Rodriguez DV. Effectiveness of topical insulin for the treatment of surface corneal pathologies. Arch Soc Esp Oftalmol (Engl Ed). 2023 Apr;98(4):220-232. doi: 10.1016/j.oftale.2023.03.007. Epub 2023 Mar 5. PMID 36871851
- [Background] Stuard WL, Titone R, Robertson DM. The IGF/Insulin-IGFBP Axis in Corneal Development, Wound Healing, and Disease. Front Endocrinol (Lausanne). 2020 Mar 3;11:24. doi: 10.3389/fendo.2020.00024. eCollection 2020. PMID 32194500